CLINICAL TRIAL: NCT05105919
Title: Assessing Pharmacokinetics and Pharmacodynamics of Daily Enteric-coated Aspirin in Patients With StablE Diabetes: APPEASED Study Phase 1
Brief Title: Assessing Pharmacokinetics and Pharmacodynamics of Daily Enteric-coated Aspirin in Patients With StablE Diabetes
Acronym: APPEASED
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Montreal Heart Institute (Other)
Collaborators: Institut de Recherches Cliniques de Montreal (Other)
Responsible Party: Principal Investigator, Guillaume Marquis-Gravel, Interventional Cardiologist, Associate Professor of Medicine, Montreal Heart Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ICM 2021-2919
Record Dates: First submitted 2021-10-23; First posted 2021-11-03 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes; Aspirin; Acetylsalicylic acid; Pharmacodynamics
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Aspirin

STUDY DESIGN:
Intervention Model Description: This is a single arm open-label feasibility phase 1 trial. The aim of the study if to determine the number of potentially eligible participants and the monthly recruitment rate at the MHI (Montreal Heart Institute), the Centre Épic and the IRCM (Institut de recherche clinique de Montréal) as well as participants adherence to study protocol to determine feasibility of a phase 2 trial within these centers.
Masking Description: All enrolled participants will receive the same treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Aspirin therapy (Experimental): All participants will be assigned to aspirin therapy. Participants will receive 80 mg of enteric coated aspirin per day for a 7 day period.
  Interventions: Drug: Aspirin 80 mg EC Tab

INTERVENTIONS:
Drug: Aspirin 80 mg EC Tab — Participants will receive a 7 day supply of Aspirin 80 mg EC Tab and will be instructed to take the drug at the same time every day for 7 days.

SUMMARY:
This phase 1 study will include patients suffering from type 2 diabetes mellitus and will study their response to enteric coated aspirin at a dose of 80 mg per day for a 7-day period. The aims are to determine the feasibility of a phase 2 larger scale trial, and to characterize the prevalence of incomplete platelet inhibition after exposure to EC aspirin at doses of 80 mg once daily. Platelet function will be assessed at baseline and a day 7.

DETAILED DESCRIPTION:
APPEASED is a phase 1 open-label single arm pilot trial, aiming to determine the feasibility of a larger confirmatory randomized trial, and to characterize the prevalence of incomplete platelet inhibition after exposure to EC aspirin at doses of 80 mg once daily in patients with type 2 diabetes. The primary endpoint will be incomplete platelet aggregation in response to arachidonic acid at a concentration of 1mM, measured by LTA (Light Transmission Agregometry). For every platelet function assessment, serum salicylate concentration will also be measured. Upon the screening visit (day 0), blood will be drawn and baseline platelet function will be assessed. A 7 day supply of aspirin will be given to participants meeting the eligibility criteria. Participants will be instructed to take 1 dose of 80 mg of enteric coated aspirin per day at the same time every day. Upon day 7, participants will return for a second visit before the intake of their daily aspirin, and therefore 24 hours after the previous dose of aspirin was taken. Blood will be drawn and platelet function will be assessed in the same manner as described previously. Participants will then take their final dose of aspirin under supervision, and a final blood sample will be collected and platelet function will be assessed two hours later.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years;
2. Participant must be naïve to aspirin, defined as absence of chronic treatment with aspirin within the previous 3 months, and of any aspirin use within the previous 2 weeks;
3. Type 2 diabetes, based on at least one of the following criteria: (5)

   * Chronic treatment with oral antihyperglycemic agents or insulin therapy;
   * Fasting Plasma Glucose (FPG) ≥ 126 mg/dL (7.0 mmol/L) (fasting is defined as no caloric intake for at least 8h);
   * 2-h Plasma Glucose (2h-PG) ≥200 mg/dL (11.1 mmol/L) during the oral glucose tolerance test (OGTT);
   * A1C ≥ 6.5% (48 mmol/mol);
4. Willing to attend all study visits.

Exclusion Criteria:

1. Definitive indication for aspirin, including any evidence of atherosclerotic disease, previous or current;
2. Known hypersensitivity to aspirin;
3. High-risk GI bleeding features, such as known H. pylori infection, past or present ulcer, history of bleeding from the GI tract;
4. Bleeding diathesis;
5. History of hematological malignancy or myelodysplasia;
6. Platelet count or hemoglobin levels outside of the normal reference range;
7. Planned major surgical procedure within 30 days of enrolment;
8. Chronic inflammatory disease requiring regular anti-inflammatory treatment;
9. Chronic treatment with an oral anticoagulant, an antiplatelet agent, NSAIDs or systemic steroids;
10. Active cancer;
11. Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-08-26 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Incomplete platelet aggregation inhibition by aspirin at 7 days. | 7 days.
  Incomplete platelet aggregation inhibition will be defined as ≥ 20% of residual platelet aggregation in response to arachidonic acid at a concentration of 1mM, measured by LTA (Light Transmission Aggregometry).

SECONDARY OUTCOMES:
Serum levels of thromboxane B2 | 7 days.
  Serum levels of thromboxane B2, measured by immunoassay > 3.1 ng/ml will be considered as evidence of recovery of platelet function.
Platelet aggregation response to various agonists | 7 days.
  Platelet reactivity to various agonists such as ADP (Adenosine Diphosphate), TRAP (Thrombin receptor activating peptide), epinephrine and collagen will be assessed by LTA (Light Transmission Agregometry).

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Marquis-Gravel, MD, MSc, Principal Investigator — Montreal Heart Institute
Locations (1):
- Montreal Heart Institute, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Marquis-Gravel G, Roe MT, Harrington RA, Munoz D, Hernandez AF, Jones WS. Revisiting the Role of Aspirin for the Primary Prevention of Cardiovascular Disease. Circulation. 2019 Sep 24;140(13):1115-1124. doi: 10.1161/CIRCULATIONAHA.119.040205. Epub 2019 Sep 23. PMID 31545683
- [Result] ASCEND Study Collaborative Group; Bowman L, Mafham M, Wallendszus K, Stevens W, Buck G, Barton J, Murphy K, Aung T, Haynes R, Cox J, Murawska A, Young A, Lay M, Chen F, Sammons E, Waters E, Adler A, Bodansky J, Farmer A, McPherson R, Neil A, Simpson D, Peto R, Baigent C, Collins R, Parish S, Armitage J. Effects of Aspirin for Primary Prevention in Persons with Diabetes Mellitus. N Engl J Med. 2018 Oct 18;379(16):1529-1539. doi: 10.1056/NEJMoa1804988. Epub 2018 Aug 26. PMID 30146931
- [Result] Lordkipanidze M, Pharand C, Schampaert E, Palisaitis DA, Diodati JG. Heterogeneity in platelet cyclooxygenase inhibition by aspirin in coronary artery disease. Int J Cardiol. 2011 Jul 1;150(1):39-44. doi: 10.1016/j.ijcard.2010.02.025. Epub 2010 Mar 7. PMID 20207433
- [Result] Bhatt DL, Grosser T, Dong JF, Logan D, Jeske W, Angiolillo DJ, Frelinger AL 3rd, Lei L, Liang J, Moore JE, Cryer B, Marathi U. Enteric Coating and Aspirin Nonresponsiveness in Patients With Type 2 Diabetes Mellitus. J Am Coll Cardiol. 2017 Feb 14;69(6):603-612. doi: 10.1016/j.jacc.2016.11.050. Epub 2017 Jan 11. PMID 28089180